CLINICAL TRIAL: NCT01056640
Title: A Randomized Controlled Trial of Telemonitoring Versus Usual Care in a High Risk Elderly Population.
Brief Title: Telemonitoring Versus Usual Care
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Paul Takahashi,, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-005259
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-01

CONDITIONS: Health Care Quality; Health Care Access
Keywords: telemonitoring; usual care; elderly; hospitalization; Emergency room visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Telemonitoring (Experimental): The Intel Health Guide is an FDA approved device that is placed within the patient's home and is connected to the health system via broadband internet, 3G network or phone line. This device has video monitoring which allows a real time face to face interaction with the provider. This allows for an individualized home care plan based upon multiple concerns which have not been adequately studied.
  Interventions: Device: Intel Health Guide
- Usual Care (Active Comparator): The usual care intervention will include appropriate primary care and specialty office practice visits as required. It also includes home health care, timely post-hospital outpatient visits, a nurse generated phone call progress report within one business day of hospital dismissal, and standard clinic phone triage during business hours. It also involves a 24 hour nurse triage line for questions. Patients will be informed of the general options currently available to patients including the above as well as options for care in extended hours and at Mayo Express care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Intel Health Guide — The Intel Health Guide is an FDA approved device that is placed within the patient's home and is connected to the health system via broadband internet, 3G network or phone line.
  Arms: Home Telemonitoring
Other: Usual Care — The usual care intervention will include appropriate primary care and specialty office practice visits as required.
  Arms: Usual Care

SUMMARY:
Background: Older adults with multiple chronic illnesses are at risk for worsening functional and medical status with ensuing hospitalization. One goal of medical care is to prevent this decline. One method that may help slow this functional and medical decline is home telemonitoring.

Specific aim: To determine the effectiveness of home telemonitoring compared to usual care in reducing combined outcomes of hospitalization and emergency room visits in an at risk population over 60 years of age.

Materials and Methods: This will be a randomized trial of 200 patients into one of two interventions. Home telemonitoring involves the use of a computer device at home which records biometric and symptom data from patients. This information is monitored by mid level providers associated with the primary care medical practice. Usual care involves patients who make appointments with their providers as problems arise and utilize ongoing support like a 24 hours nurse line. The study participants are adults over 60 years of age within the highest 10% on elderly risk assessment (ERA) scores. Patients will have initial evaluations of gait, quality of life (SF12), Kokmen test of mental status, and PHQ 9. Patients will be followed for 1 year for primary outcomes of hospitalizations and emergency room visits. Secondary analysis will include quality of life, compliance with the device and attitudes about telemonitoring. Sample size is based upon an 80% power to detect a 36% difference between the groups. The primary analysis will involve Cox proportional time to event analysis comparing both interventions for telemonitoring or usual care. Secondary analysis will use T-test comparisons for continuous variables (quality of life, attitudes) and chi square for proportional analysis.

ELIGIBILITY:
Inclusion:

1. at least 60 years of age;
2. have an Elder Risk Assessment (ERA) Index score of 16 or greater;
3. Are able to participate fully in all aspects of the study;
4. Have been provided with, understand, and have signed the informed consent;

Exclusion:

1. patients who are currently residing in a nursing home
2. patients with a clinical diagnosis of dementia
3. patients with a score of ≤29 on the Kokmen short test of mental status
4. patients for whom we cannot obtain informed consent.
5. patient under the age of 60 will also be excluded from participating.
6. patients who have not granted Universal Research Authorization to use medical records.
7. patients will also be excluded if the subject would not be able to use the interventional machine

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Takahashi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Takahashi PY, Pecina JL, Upatising B, Chaudhry R, Shah ND, Van Houten H, Cha S, Croghan I, Naessens JM, Hanson GJ. A randomized controlled trial of telemonitoring in older adults with multiple health issues to prevent hospitalizations and emergency department visits. Arch Intern Med. 2012 May 28;172(10):773-9. doi: 10.1001/archinternmed.2012.256. PMID 22507696
- [Derived] Takahashi PY, Hanson GJ, Pecina JL, Stroebel RJ, Chaudhry R, Shah ND, Naessens JM. A randomized controlled trial of telemonitoring in older adults with multiple chronic conditions: the Tele-ERA study. BMC Health Serv Res. 2010 Sep 1;10:255. doi: 10.1186/1472-6963-10-255. PMID 20809953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 11/21/09 and completed on 08/07/10. Interested subjects who passed a phone prescreen were seen at the study center or in their homes for consenting and additional study procedures to determine eligibility.
Pre-assignment Details: If study subjects consented to be in study and were found to be eligible, they were randomized to be in study. If they were randomized to receive the telemonitor, within 3-5 days the study team make arrangements to go to their home to install the telemonitor.
Groups:
- Home Telemonitoring: The Intel Health Guide is an FDA approved device that is placed within the patient's home and is connected to the health system via broadband internet, 3G network or phone line. This device has video monitoring which allows a real time face to face interaction with the provider. This allows for an individualized home care plan based upon multiple concerns which have not been adequately studied.
  Intel Health Guide : The Intel Health Guide is an FDA approved device that is placed within the patient's home and is connected to the health system via broadband internet, 3G network or phone line.
- Usual Care: The usual care intervention will include appropriate primary care and specialty office practice visits as required. It also includes home health care, timely post-hospital outpatient visits, a nurse generated phone call progress report within one business day of hospital dismissal, and standard clinic phone triage during business hours. It also involves a 24 hour nurse triage line for questions. Patients will be informed of the general options currently available to patients including the above as well as options for care in extended hours and at Mayo Express care.
  Usual Care : The usual care intervention will include appropriate primary care and specialty office practice visits as required.
Period: Overall Study
Arm/Group | Home Telemonitoring | Usual Care
Started | 102 | 103
Completed | 76 | 91
Not Completed | 26 | 12
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Death | 15 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Telemonitoring | Usual Care | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 97 | 100 | 197
Age Continuous [Mean (Standard Deviation); unit: years] | 80.3 (8.9) | 80.2 (7.6) | 80.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 59 | 111
  Male | 50 | 44 | 94

OUTCOME MEASURES:

1. Primary Outcome: Mean # Participants Who Had Hospitalizations or ED Visits Compared to Usual Care in a High Risk Group of Adults ≥ 60 Years of Age With Mixed Chronic Disease.
Time Frame: 12 months
Population: This study utilized an intent-to-treat method. Everyone randomized to study was included in the analysis
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Home Telemonitoring | Usual Care
Number analyzed (Participants) | 102 | 103
hospitalizations | 65 (63.7) | 59 (57.3)
Statistical Analysis 1: Comparison: Home Telemonitoring vs Usual Care; All analyses were performed using an intent-to-treat method. Wilcoxon rank sum test, 2-sample t test, or Chi-Square analysis was used to compare baseline characteristics. The primary end points of combined and individual percentages of hospitalizations and ED visits were compared using Chi-Square test. Statistical adjustment was planned only if there were statistical differences in clinical variables between the groups. All tests for significance used a 2-sided P value of .05; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon Rank Sum test, 2-sample t-test and Chi-square analysis were all used; Odds Ratio (OR) = 1.310, 95% CI 2-sided [0.747 to 2.297], Standard Error of Mean 0.2865

ADVERSE EVENTS:
Arm/Group | Home Telemonitoring | Usual Care
Serious Adverse Events (participants affected / at risk) | 15/102 | 4/103
Other Adverse Events (participants affected / at risk) | 0/102 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Telemonitoring (N=102) | Usual Care (N=103)
Death (Social circumstances) | 15 (15) | 4 (4)

LIMITATIONS AND CAVEATS:
Patients in the usual care group had access to a tertiary care hospital and to some case management for treatment of heart failure and diabetes. These services may have biased the results to show no difference between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes